CLINICAL TRIAL: NCT04849845
Title: DOS [Dosing Optimization Study]: Open-label, Single-arm, Proof-of-Concept Dosing Study of Afrezza® in Adult Subjects 18 Years and Older With Type 1 or Type 2 Diabetes Mellitus
Brief Title: Afrezza® Dosing Optimization Study
Acronym: DOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-191
Record Dates: First submitted 2021-04-16; First posted 2021-04-19 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Afrezza; Dosing; Technosphere; Inhaled; Insulin; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Insulin Resistance; Respiratory Aspiration; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Afrezza (Experimental): The test product is defined as Afrezza [insulin human] inhalation powder administered using the Afrezza inhaler. In addition, subjects will take their personal basal insulin while enrolled in the study.
  Interventions: Combination Product: Afrezza Dose 1; Combination Product: Afrezza Dose 2

INTERVENTIONS:
Combination Product: Afrezza Dose 1 — The first dose of Afrezza will be based on the dose of subcutaneous rapid-acting analogue (RAA) insulin that the subject would normally take for the standardized meal, converted according to the guidelines provided in the current Afrezza U.S. prescribing information.
Combination Product: Afrezza Dose 2 — The second dose of Afrezza will be based on the dose of subcutaneous rapid-acting analogue that the subject would normally take for the standardized meal, converted by multiplying their RAA dose by 2 and rounding down to the nearest Afrezza cartridge size.

SUMMARY:
MKC-TI-191 is a Phase 4, single-arm, multicenter, proof-of-concept clinical trial evaluating the efficacy and safety of Afrezza, administered according to the current Afrezza prescribing information (PI) compared to a titrated dose, in combination with a basal insulin in adult subjects (≥18 years of age) with type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM). Eligible subjects will be on a stable regimen consisting of a basal bolus insulin therapy prior to screening. The study is composed of up to 4 clinic visits (screening, 2 treatment visits, and a follow-up visit). Two individual doses of Afrezza will be administered during a meal challenge at Visits 2 and 3. The duration of each subject's participation in the trial is expected to be approximately 2 weeks.

DETAILED DESCRIPTION:
Screening (Visit 1): Informed consent and California Experimental Subjects Bill of Rights will be signed and eligibility confirmed. Eligible subjects will be enrolled at Visit 1.

Subjects will come into the clinic in a fasting state for a meal challenge and individual dose of Afrezza during Visits 2 and 3. At the beginning of each visit, before their dose of Afrezza, subjects will have FEV1 measurements taken in the clinic. Each meal challenge will consist of 1 to 2 bottles of nutritional shake to be fully consumed within 15 minutes. The nutritional shake will contain approximately 240 calories, 41 g carbohydrate, 10 g protein, and 4 g fat per bottle. Each Afrezza dose will be administered at the start of the meal challenge.

Visit 2: The first dose of Afrezza will be based on the dose of subcutaneous (SC) rapid-acting analogue (RAA) insulin that the subject would normally take, converted according to the guidelines provided in the current Afrezza prescribing information. If subject's normal RAA dose is <4 units or 5 units, subject will be asked to consume enough nutritional shake, per their normal I:C ratio, to cover an RAA dose of 4 units or ≥6 units such that their Afrezza dose at Visit 3 is higher than the dose taken at Visit 2. After completing the standardized meal challenge, the Investigator will decide, based on the subject's glucose excursion at Visit 2, if the subject should proceed to Visit 3 where a second dose of Afrezza will be administered.

Visit 3: The second dose of Afrezza will be based on the dose of SC RAA that the subject would normally take, converted by multiplying their RAA dose by 2 and rounding down to the nearest Afrezza cartridge size.

Follow-up Visit (Visit 4): Subjects will return for safety assessments, including a final FEV1 measurement, 24 to 72 hours after their last dose of Afrezza.

ELIGIBILITY:
Subjects will be asked to provide a recent negative COVID-19 test (if available), confirm they have no symptoms of COVID-19, or provide evidence of COVID-19 vaccination.

Inclusion Criteria:

1. Subjects ≥18 years of age at the time of signing the informed consent form
2. Clinical diagnosis of T1DM or T2DM (per the Investigator) and on a stable basal-bolus insulin regimen

Exclusion Criteria:

1. History of asthma, chronic obstructive pulmonary disease, or any other clinically important pulmonary disease (e.g., cystic fibrosis, bronchopulmonary dysplasia), use of any medications to treat such conditions within the last year, or significant congenital or acquired cardiopulmonary disease
2. History of serious complications of diabetes (e.g., active proliferative retinopathy or symptomatic autonomic neuropathy)
3. On dialysis
4. Respiratory tract infection within 14 days before screening (subject may return 14 days after resolution of symptoms for rescreening)
5. Treatment with any investigational drug in the past 30 days or an investigational device in the past 2 weeks
6. Any disease other than diabetes or initiation of any new medication that, in the judgment of the Investigator, could have a direct impact on glycemic control during the study
7. Use of antiadrenergic drugs (e.g., beta blockers and clonidine)
8. Any concurrent illness (other than diabetes mellitus) not controlled by a stable therapeutic regimen
9. History of a significant eating disorder (e.g., anorexia or bulimia nervosa)
10. Current drug or alcohol abuse or a history of drug or alcohol abuse that, in the opinion of the Investigator or the Sponsor, would make the subject an unsuitable candidate for participation in the study
11. History of smoking (includes cigarettes, cigars, pipes, vaping devices, and marijuana) in the 6 months before screening
12. Female subject who is pregnant, breastfeeding, intends to become pregnant, or is of child-bearing potential and not using adequate contraceptive methods as required by local regulation or practice (may include sexual abstinence)
13. An event of severe hypoglycemia, as judged by the Investigator, within the 90 days before screening
14. An episode of diabetic ketoacidosis (DKA) requiring hospitalization within the 90 days before screening
15. Exposure to Afrezza in the 30 days before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kaiserman, MD, Study Director — Mannkind Corporation
Locations (2):
- United States (2):
  - AMCR Institute, Escondido, California
  - Diablo Clinical Research, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2021 and May 2021, a total of 20 subjects were enrolled at two investigational sites in the US.
Groups:
- Afrezza: The test product was defined as Afrezza [insulin human] inhalation powder administered using the Afrezza inhaler. In addition, subjects took their personal basal insulin while enrolled in the study.
  The first dose of Afrezza was based on the dose of subcutaneous rapid-acting analogue (RAA) insulin that the subject would normally take for the standardized meal, converted according to the guidelines provided in the current Afrezza U.S. prescribing information.
  The second dose of Afrezza was based on the dose of subcutaneous rapid-acting analogue that the subject would normally take for the standardized meal, converted by multiplying their RAA dose by 2 and rounding down to the nearest Afrezza cartridge size.
Period: Afrezza Dose 1
Arm/Group | Afrezza
Started | 20
Completed | 20
Not Completed | 0
Period: Afrezza Dose 2
Arm/Group | Afrezza
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Afrezza: The test product was defined as Afrezza [insulin human] inhalation powder administered using the Afrezza inhaler. In addition, subjects took their personal basal insulin while enrolled in the study.
  Afrezza Dose 1: The first dose of Afrezza was based on the dose of subcutaneous rapid-acting analogue (RAA) insulin that the subject would normally take for the standardized meal, converted according to the guidelines provided in the current Afrezza U.S. prescribing information.
  Afrezza Dose 2: The second dose of Afrezza was based on the dose of subcutaneous rapid-acting analogue that the subject would normally take for the standardized meal, converted by multiplying their RAA dose by 2 and rounding down to the nearest Afrezza cartridge size.
Arm/Group | Afrezza
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (13.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 20
HbA1c [Mean (Standard Deviation); unit: percentage of Hemoglobin A1c] — Hemoglobin A1C
  percentage of Hemoglobin A1c | 6.66 (0.84)
Diabetes type [Count of Participants; unit: Participants]
  Type 1 diabetes | 18
  Type 2 diabetes | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index
  kg/m^2 | 26.9 (6.97)

OUTCOME MEASURES:

1. Primary Outcome: Post-prandial Glucose Excursion
Description: Mean glucose change from baseline (or postprandial glucose excursion [PPGE]) based on self-monitored blood glucose (SMBG) at 15, 30, 45, 60, 90 and 120 minutes after the dose of Afrezza with baseline defined as SMBG at the time of the dose of Afrezza (t=0)
Time Frame: 120 minutes post-dose
Population: Intent to treat, including all subjects in the safety population, had a baseline value and at least one postbaseline value
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Afrezza Dose 1: The test product was defined as Afrezza [insulin human] inhalation powder administered using the Afrezza inhaler. In addition, subjects took their personal basal insulin while enrolled in the study.
  The first dose of Afrezza was based on the dose of subcutaneous rapid-acting analogue (RAA) insulin that the subject would normally take for the standardized meal, converted according to the guidelines provided in the current Afrezza U.S. prescribing information.
- Afrezza Dose 2: The test product was defined as Afrezza [insulin human] inhalation powder administered using the Afrezza inhaler. In addition, subjects took their personal basal insulin while enrolled in the study.
  The second dose of Afrezza was based on the dose of subcutaneous rapid-acting analogue that the subject would normally take for the standardized meal, converted by multiplying their RAA dose by 2 and rounding down to the nearest Afrezza cartridge size.
Arm/Group | Afrezza Dose 1 | Afrezza Dose 2
Number analyzed (Participants) | 20 | 20
mg/dL
  15 minutes PPGE | 6.8 (3.3) | 5.6 (2.5)
  30 minutes PPGE | 25.9 (5.7) | 21.9 (5.6)
  45 minutes PPGE | 48.9 (6.9) | 27.0 (6.6)
  60 minutes PPGE | 64.2 (7.9) | 34.3 (8.1)
  90 minutes PPGE | 82.8 (14.3) | 36.0 (10.2)
  120 minutes PPGE | 88.6 (17.7) | 36.9 (13.1)

2. Secondary Outcome: Number of Subjects With at Least 1 Event of Level 1 Hypoglycemia
Description: Number of subjects with at least 1 event (also referred to as incidence) of Level 1 hypoglycemia (<70mg/dL) within the 120 minutes after Afrezza dosing as confirmed by SMBG.
Time Frame: 120 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Afrezza Dose 1 | Afrezza Dose 2
Number analyzed (Participants) | 20 | 20
Participants | 0 | 1

3. Secondary Outcome: Percent of Level 1 Hypoglycemia
Description: Percent of total SMBG measurements <70 mg/dL (Level 1 hypoglycemia) within the 120 minutes after Afrezza dosing.
Time Frame: 120 minutes
Population: as for outcome 1
Measure: Number; unit: SMBG Measurements
Units Other Than Participants: SMBG Measurements
Arm/Group | Afrezza Dose 1 | Afrezza Dose 2
Number analyzed (Participants) | 20 | 20
Number analyzed (SMBG Measurements) | 120 | 120
SMBG Measurements | 0 | 2

4. Secondary Outcome: Number of Subjects With at Least 1 Event of Level 2 Hypoglycemia
Description: Number of subjects with at least 1 event (also referred to as incidence) of Level 2 hypoglycemia (<54mg/dL) within the 120 minutes after Afrezza dosing as confirmed by SMBG.
Time Frame: 120 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Afrezza Dose 1 | Afrezza Dose 2
Number analyzed (Participants) | 20 | 20
Participants | 0 | 1

5. Secondary Outcome: Percent of Level 2 Hypoglycemia
Description: Percent of total SMBG measurements <54 mg/dL (Level 2 hypoglycemia) within the 120 minutes after Afrezza dosing
Time Frame: 120 minutes
Population: as for outcome 1
Measure: Number; unit: SMBG Measurements
Units Other Than Participants: SMBG Measurements
Arm/Group | Afrezza Dose 1 | Afrezza Dose 2
Number analyzed (Participants) | 20 | 20
Number analyzed (SMBG Measurements) | 120 | 120
SMBG Measurements | 0 | 1

6. Secondary Outcome: Number of Subjects With At Least 1 Event of Severe Hypoglycemia
Description: Number of subjects with at least 1 event (also referred to as incidence) of severe hypoglycemia, defined as events requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions within the 120 minutes after Afrezza dosing.
Time Frame: 120 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Afrezza Dose 1 | Afrezza Dose 2
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

7. Secondary Outcome: Change in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Between Two Points, Baseline and 120 Minutes Post-Afrezza Dose
Description: Change in percent predicted forced expiratory volume in 1 second (FEV1) between two points (value at 120 minutes post-Afrezza dose minus value at baseline). Standard deviation was not reported.
Time Frame: 120 minutes post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in percent predicted FEV1
Arm/Group | Afrezza Dose 1 | Afrezza Dose 2
Number analyzed (Participants) | 20 | 20
change in percent predicted FEV1 | 0.63 (8.25) | -2.55 (5.78)

ADVERSE EVENTS:
Time Frame: Duration of the two treatment visits (~8 hours)
Arm/Group | Afrezza Dose 1 | Afrezza Dose 2
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Afrezza Dose 1 (N=20) | Afrezza Dose 2 (N=20)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
DOS had no planned or conducted hypothesis testing, and no alpha adjustment was made to account for multiple testing of exploratory endpoints. Instead, DOS aimed to be a small-scale test of the higher dose suggested by previous studies and clinical experience. With no formal hypothesis testing, descriptive statistical comparisons are used to assess the efficacy and safety outcomes of the higher dose for purposes of generating hypothesis for a larger study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose any of the results arising out of or in connection with the clinical trial without the prior express written consent of the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT04849845/Prot_SAP_001.pdf